CLINICAL TRIAL: NCT06194708
Title: Reasons for Non-reversal of Temporary Stomas After Surgeries of Mid-low Rectal Cancer （NORESTO Study）on Behalf of Chinese Ostomy Collaboration Group (COCG-02)
Brief Title: Reasons for Non-reversal of Temporary Stomas After Surgeries of Mid-low Rectal Cancer （NORESTO Study）
Status: Recruiting | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: COCG-02
Record Dates: First submitted 2023-12-22; First posted 2024-01-08 (Actual); Last update posted 2024-01-08 (Actual); Status verified 2023-01

CONDITIONS: Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Mid-low rectal cancer patients with temporary stoma after radical surgery

SUMMARY:
The goal of this observational study is to learn about in mid-low rectal patients who received temporary ostomies after surgery of the primary tumors. The main questions it aims to answer are:

* To explore the proportion of temporary stomas that cannot be reversed after radical surgery for mid-low rectal cancer and their main causes.
* To use the basic information we collected from patients before and during surgery to develop an individualized model for predicting the time of stoma reversal and explore the risk factors affecting stoma reversal.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed as rectal adenocarcinoma;
* The tumor is located within 12cm from the anal verge;
* Primary tumor is radically resected;
* The patient received a temporary ostomy during the in-hospital visit of the resection of the primary tumor.

Exclusion Criteria:

* The stoma was initially recognized as permanent stoma;
* Patients with distant metastasis;
* Patients with multi-primary colorectal cancer.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In-hospital rectal cancer patients who underwent radical resection of the primary lesion
Sampling Method: Probability Sample
Enrollment: 235 (Estimated)
Dates: Start 2023-05-15 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
1-year non-reversal rate of temporary stoma | 1 year after ostomy

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No